CLINICAL TRIAL: NCT04014751
Title: Expansion, Implementation & Evaluation of Electronic Health Record (EHR)-Integrated Patient-Reported Symptom Screening in a Multi-Site Cancer Center
Brief Title: Evaluation of a Symptom and Needs Assessment for Patients With Cancer
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sofia Garcia, Research Associate Professor, Northwestern University
Other Study IDs: 1R18HS026170-01 (AHRQ)
Record Dates: First submitted 2019-06-04; First posted 2019-07-10 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Cancer
Keywords: Symptom-monitoring
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Symptom Monitoring Cohort: This cohort will include up to1,050 cancer patients being seen at regional Northwestern Medicine (NM) cancer centers for their cancer care. Patients who have recently completed an on-line, EHR-integrated patient-reported symptom and needs assessment as part of their regular care will be invited to complete a survey at baseline, 6- and 12-months targeting the assessment of their symptoms, healthcare experiences and utilization. Patients may also be invited to participate in a one-time interview or focus group designed to help study investigators better understand the value of the symptom and needs assessment from the patient perspective.
  Interventions: Other: Symptom Monitoring Intervention

INTERVENTIONS:
Other: Symptom Monitoring Intervention — This study involves a cancer care delivery process improvement component where all cohort participants, at specified timepoints, are assessed for psychological distress, pain, fatigue, physical function, practical and supportive needs, and dietary and nutritional needs. Patients with severe elevations in psychological distress, physical symptoms or those who endorse supportive care and/or dietary needs are triaged in real time to appropriate providers within the health system (i.e., social work, nursing pool, nutrition services) to address elevated scores and/or stated needs. As such, within the context of this process improvement care delivery project, real time referrals function as interventional processes within the health system to route patients to relevant points of care based on their needs.

SUMMARY:
This is a quality improvement study that aims to improve on the timely identification and management of symptoms and supportive care needs in patients with cancer. The study will be evaluating the relative success of an existing on-line patient-reported symptom and needs assessment, and then the implementation and use of an updated version of the symptom and needs assessment with Northwestern Medicine (NM) cancer patients. It also aims to evaluate the impact of the symptom and needs assessment system on healthcare delivery and quality of care. Participants who complete the symptom and needs assessment as part of their usual care are invited to participate in the study by agreeing to complete an on-line survey (at 3 different time points) that asks about quality of life, adverse symptoms related to cancer and cancer treatment, patient experiences with their cancer care team, and the healthcare services they have received. Patients may also be invited to participate in a one-time interview or focus group about patient experiences with the symptom and needs assessment.

DETAILED DESCRIPTION:
Cancer patients' under-identified symptoms and concerns can result in treatment interference, poor care satisfaction, compromised health-related quality of life, and taxed healthcare systems. Cancer care organizations have emphasized the need for symptom assessment and management within quality cancer care delivery. We have leveraged health information technology to pilot and implement the Lurie Screening Initiative in the Robert H. Lurie Comprehensive Cancer Center (RHLCCC) within the Central region of Northwestern Medicine (NM). Following two pilot implementation projects, the screening initiative program is live in RHLCCC clinics. It allows patients to complete Patient Reported Outcomes Measurement Information System computer adaptive tests (PROMIS CATs) assessing depression, anxiety, fatigue, pain, and physical function, along with checklists of supportive care needs, within the electronic health record (EHR). Patients can do so at home via MyChart (a patient portal of their EHR) or in clinic via an EHR hyperlink. Assessment results immediately populate the EHR; severe symptoms and endorsed supportive care needs trigger notifications to clinicians (social workers, dieticians, oncologists & oncology nurses) who can then make referrals and care decisions in real time.

This study will expand and evaluate implementation of the screening initiative via these aims:

Aim 1. Evaluate the impact of system-wide implementation of the program on patient and system outcomes over 12 months via (a) a quality improvement study (estimated n=4,000 cases) to compare the impact of the program (versus usual care) on EHR-documented health care usage and patient satisfaction using a stepped wedge design in which clusters of study sites will gradually be assigned to cross from serving as a control to implementing the program and (b) a human subjects substudy (n=1,000) with patients who will complete the symptom monitoring and other patient-reported outcomes (PRO) measures of health care usage and satisfaction at baseline, 6 & 12 months. We will examine differences in PROs between participants whose screening responses trigger clinical alerts and those who do not. We will also explore longitudinal trajectories of PRO scores

Aim 3. Identify implementation facilitators and barriers to system-wide expansion of the program. We will conduct qualitative research to gather feedback from patients participating in the program expansion (n=50). This will include multiple assessments throughout implementation.

ELIGIBILITY:
1. Must have medical chart confirmed diagnosis of a solid or hematological malignancy
2. Must have had oncology services at a Northwestern Medicine location within the past 12 months
3. Must have completed the current symptom monitoring assessment offered by Northwestern Medicine
4. Must be willing to complete electronic patient-reported measures (i.e. patient reported health care utilization and satisfaction surveys) at baseline, 6-month, and 12-month follow-up time points, and
5. Must consent to give authorized study staff access to details of their cancer diagnosis and treatment as documented in their electronic health record
6. If participating in a semi-structured interview or focus group, must consent to have their comments audio-recorded

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients at Northwestern Medicine (NM) who have a confirmed diagnosis of a solid or hematological malignancy and have had oncology services at NM within the past 12-months.
Sampling Method: Non-Probability Sample
Enrollment: 1166 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Effects of the symptom monitoring system on patient-reported quality of life related to cancer and cancer treatment | Change from baseline quality of life at 12-months
  Quality of life will be assessed using a brief, validated 7-item patient-reported questionnaire (Functional Assessment of Cancer Therapy-General 7-item or FACT-G7) that asks about symptoms of fatigue, pain, and nausea, sleep quality and contentment with life.
Effects of the symptom monitoring system on severity of patient-reported symptoms related to cancer and cancer treatment | Change from baseline symptom severity at 12-months
  Symptom severity will be assessed via a Patient-Reported Outcome Measurement Information System (PROMIS) computer adaptive test (CAT) that will ask about depression, anxiety, pain, fatigue, and physical functioning. CAT items are dynamically selected for administration from an item bank based upon the respondent's previous answers. Patient usually completes 4-12 items with a high level of measurement.
Effects of the symptom monitoring system on patient-reported adverse events related to cancer and cancer treatment | Change from baseline adverse events at 12-months
  Adverse events will be assessed using the Patient-Reported Outcomes- Common Terminology Criteria for Adverse Events (PRO-CTCAE™) assessment. The PRO-CTCAE questionnaire will ask questions about nausea, constipation, insomnia, vomiting, and diarrhea.
Impact of the symptom monitoring system on health care services used by patients | Change from baseline use of healthcare services at 12 months
  Utilization of services related to physical and mental health will be measured using a patient-reported questionnaire to assess healthcare services used by participants, such as number of emergency room visits, oncology urgent care visits, general urgent care visits, doctor visits, referrals for services within and outside the health system, and overnight stays in the hospital.

SECONDARY OUTCOMES:
Impact of the symptom monitoring system on patient experiences with their cancer care team | Change from baseline patient experiences with their cancer care team at 12 months
  Patient experiences with their cancer care team will be measured using components of a standardized measure (Consumer Assessment of Healthcare Providers and Systems or CAHPS) designed to assess patient experiences with their healthcare provider and system.
Patient experiences (barriers and facilitators) using the symptom and needs assessment | Patient experiences will be assessed at one time point between baseline and 12 months
  Patient experiences with the symptom and needs assessment will be evaluated using qualitative methods (semi-structured interview or focus group)

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Garcia, PHD, Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith JD, Merle JL, Webster KA, Cahue S, Penedo FJ, Garcia SF. Tracking dynamic changes in implementation strategies over time within a hybrid type 2 trial of an electronic patient-reported oncology symptom and needs monitoring program. Front Health Serv. 2022 Nov 1;2:983217. doi: 10.3389/frhs.2022.983217. eCollection 2022. PMID 36925901
- [Derived] Garcia SF, Smith JD, Kallen M, Webster KA, Lyleroehr M, Kircher S, Bass M, Cella D, Penedo FJ. Protocol for a type 2 hybrid effectiveness-implementation study expanding, implementing and evaluating electronic health record-integrated patient-reported symptom monitoring in a multisite cancer centre. BMJ Open. 2022 May 3;12(5):e059563. doi: 10.1136/bmjopen-2021-059563. PMID 35504641